CLINICAL TRIAL: NCT02486068
Title: ABSORB Bioresorbable Scaffold vs. Xience Metallic Stent for Prevention of Restenosis Following Percutaneous Coronary Intervention in Patients at High Risk of Restenosis
Brief Title: ABSORB Bioresorbable Scaffold vs. Xience Metallic Stent for Prevention of Restenosis in Patients at High Risk of Restenosis
Acronym: Compare Absorb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPARE ABSORB
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABSORB scaffold (Experimental): Patient will undergoes elective or emergent percutaneous coronary intervention and will be treated with ABSORB scaffold.
  Interventions: Device: ABSORB scaffold
- Xience (Active Comparator): Patient will undergoes elective or emergent percutaneous coronary intervention and will be treated with Xience Prime.
  Interventions: Device: Xience

INTERVENTIONS:
Device: ABSORB scaffold
  Arms: ABSORB scaffold
Device: Xience
  Arms: Xience

SUMMARY:
The primary objectives of this trial are:

In patients at high-risk for restenosis,

* To assess non-inferiority of the everolimus-eluting bioresorbable scaffold (BRS) to the everolimus eluting cobalt chromium metallic stent (EES) in target lesion failure (TLF) at 1 year
* To assess superiority of the BRS to the EES in TLF between 3 and 7 years

ELIGIBILITY:
Inclusion Criteria:

Patients (18-75 years old) with at least one of the followings:

* High-risk characteristics for restenosis

  * Medically treated Diabetes (oral medication or insulin)
  * Multivessel disease of which more than one de-novo target lesion to be treated with the study scaffold/stent
* Complex target lesion

  * Single de-novo target lesion satisfying at least one of the following:
  * Lesion length >28 mm
  * Small vessels: Target lesion reference vessel diameter between ≥2.5 mm and ≤2.75mm
  * Lesion with pre-existing total occlusion (pre-procedural TIMI = 0)
  * Bifurcation with single stent strategy

Exclusion Criteria:

* Patients are excluded from this study if they have:
* Age <18 years or >75 years
* Known comorbidities which make patients unable to complete 7-years follow-up
* Female of childbearing potential (and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy
* Pregnant woman
* Breastfeeding woman
* Known intolerance to aspirin, heparin, PLLA, everolimus, contrast material
* Cardiogenic Shock (Killip >2)
* PCI with implantation of stents/scaffolds within previous 30 days.
* Active bleeding or coagulopathy or patients at chronic anticoagulation therapy
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint
* Renal insufficiency (GFR <45 ml/min)
* Life expectancy < 7 years
* Known non-adherence to DAPT
* Patients on oral anticoagulation therapy (including novel oral anticoagulant such as dabigatran, rivaroxaban, apixaban and edoxaban)
* LVEF <30%
* Patients at high bleeding risk who are not suitable for long-term DAPT
* Following lesion characteristics:

  * Target lesion reference vessel diameter (RVD) < 2.5 and > 4 mm
  * STEMI with RVD of >3.5mm of the culprit target lesion
  * Target lesion with in-stent/scaffold thrombosis
  * Graft lesions as target lesions
  * Aorto-ostial lesion(s)
  * Left main lesion
  * Severe tortuosity of target vessel
  * In-scaffold restenosis
  * Bifurcation target lesion with intended 2 stent/scaffold strategy
* Non-target lesion and target lesion in the same epicardial coronary artery (right coronary artery, left circumflex artery or left anterior descending artery)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1670 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2018-08-28 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
non-inferiority of the everolimus-eluting bioresorbable scaffold (Absorb) to the everolimus eluting cobalt chromium metallic stent (Xience) in target lesion failure (TLF) | 1 year
  Composite of:
  * Cardiac death
  * Myocardial infarction (MI) in target vessel territory (SCAI consensus for periprocedural MI, 3rd universal definition for spontaneous or other MI)
  * Clinically Indicated Target lesion revascularization

SECONDARY OUTCOMES:
superiority of the Absorb to the Xience in TLF between 3 and 7 years | 5 years
Superiority of the Absorb to the Xience in TLF at 7 years | 7 years
Superiority of the Absorb to the XIence in cumulative angina rate at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Smits, MD, Principal Investigator — Maastad hospital
Locations (44):
- Belgium (3):
  - Cardiovascular Center Aalst OLV, Aalst
  - CHR Citadelle, Leuven
  - UZ Leuven, Leuven
- Czechia (3):
  - University Hospital Brno, Brno
  - Cardiocentre, University Hospital Kralovske, Prague
  - Central Military Hospital, Prague
- France (5):
  - Clinique Rhône Durance, Avignon
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Privé Jacques Cartier, Massy
  - Clinique Saint-Hilaire, Rouen
  - Clinique Pasteur, Toulouse
- Germany (9):
  - Segeberger Kliniken, Bad Segeberg
  - Charité Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Elisabethkrankenhaus Essen, Essen
  - Universitätsklinikum Gießen, Giessen
  - Universität Leipzig - Herzzentrum, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Klinikum der Universität München, München
- Italy (8):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Brotzu, Cagliari
  - Ospedale San Giacomo, Castelfranco Veneto
  - Università degli studi Magna Graecia, Catanzaro
  - Università degli Studi di Napoli Federico II, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Arnas Civico Palermo, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - Catherina Ziekenhuis, Eindhoven
  - Erasmus Medisch Centrum, Rotterdam
  - Maasstadziekenhuis, Rotterdam
- Poland (4):
  - American Heart of Poland, Chrzanów
  - University Hospital Krakow, Krakow
  - Miedziowe Centrum Zdrowia SA, Lubin
  - American Heart of Poland, Tychy
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
- United Kingdom (3):
  - Royal Bournemouth Hospital, Bournemouth
  - Papworth Hospital, Cambridge
  - Freeman Hospital, Newcastle

REFERENCES:
- [Derived] Chang CC, Onuma Y, Achenbach S, Barbato E, Chevalier B, Cook S, Dudek D, Escaned J, Gori T, Kocka V, Tarantini G, West NEJ, Morice MC, Tijssen JGP, van Geuns RJ, Smits PC; COMPARE ABSORB trial investigators. Absorb Bioresorbable Scaffold Versus Xience Metallic Stent for Prevention of Restenosis Following Percutaneous Coronary Intervention in Patients at High Risk of Restenosis: Rationale and Design of the COMPARE ABSORB Trial. Cardiovasc Revasc Med. 2019 Jul;20(7):577-582. doi: 10.1016/j.carrev.2019.04.013. Epub 2019 Apr 16. PMID 31153846